CLINICAL TRIAL: NCT05252247
Title: The Effects of Immobilisation and Exercise on Homeostatic Plasticity Mechanisms in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Dennis Boye Larsen, Assistant Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20210047
Record Dates: First submitted 2022-01-19; First posted 2022-02-23 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Healthy
MeSH Terms: interventions — Immobilization; Exercise

STUDY DESIGN:
Intervention Model Description: This is a within-subject repeated measures comparisons study with one baseline session and two interventional sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conditions (Experimental): Participants will attend three sessions where two consist of immobilisation or exercise interventions.
  Interventions: Other: Immobilisation; Other: Exercise

INTERVENTIONS:
Other: Immobilisation — Eight hours prior to attending the immobilisation session, a splint will be fitted to the hand of the participant and remain until the session start.
Other: Exercise — Eight hours prior to attending the exercise session, the participant will be instructed to perform 150 ballistic finger movements every hour until the session start.

SUMMARY:
Homeostasis is important for maintaining a stable equilibrium of e.g., blood pressure, hormonal release, and release of neurotransmitters. Within the healthy brain, homeostatic plasticity mechanisms ensure stability in synaptic plasticity that maintains cortical excitability within a normal physiological range, while this regulation has been shown to be impaired in chronic pain conditions such as low back pain. Cortical excitability can also be decreased and increased experimentally, using immobilisation and exercise paradigms, respectively, yet it is unknown if this overall change in excitability is caused by a shift in homeostatic plasticity regulation. Investigating if immobilisation and exercise influences homeostatic plasticity responses, may therefore reveal important information on the malleability of homeostatic plasticity mechanisms and ways to modulate them.

DETAILED DESCRIPTION:
The aim of this study is to investigate the impact of upper limb immobilisation and physical exercise of the hand on homeostatic plasticity in healthy individuals.

The study will be performed as a randomised cross-over study where each participant take part in three sessions, separated by approximately 24 hours. During each session, the participant will answer questionnaires and undergo quantitative sensory testing (QST). Baseline measures is obtained using transcranial magnetic stimulation (TMS)-induced motor evoked potentials (MEPs), which is done before the induction of homeostatic plasticity using transcranial direct current stimulation (tDCS). MEPs are then obtained every 10 minutes for 30 minutes. Lastly, QST measures are obtained again.

As no previous studies have investigated the effect of immobilisation and exercise on homeostatic plasticity response, a sample size calculation was estimated based on MEP analysis from a previous study using α of 0.05, β of 0.80, and effect size of 0.29, yielding 22 participants. This is consistent with recent exploratory research that suggested that up to 28 participants would be needed. Therefore, the current study aimed at including 28 participants with an interim analysis performed after 10-15 inclusions.

Each participant will attend three identical experimental sessions on the same time on three consecutive days. Eight hours before attending the experimental sessions with immobilisation the participant will be fitted a splint (MANU-Hit DIGITUS POLLEX, Clinical Innovations, DK) to immobilise the right hand. Similarly, eight hours before attending the exercise session, the participant will be instructed to perform 150 ballistic finger movements with a pace of 0.5 Hz. During the experiment, the participant will be seated comfortably with arms and hands at rest. Electromyography electrodes will be placed on the right first interosseous muscle to assess the corticomotor excitability by recording of TMS induced MEPs on the left primary motor cortex. A neoprene cap will then be mounted to the head, and the optimal site for TMS (hotspot) will be identified and marked on the cap for standardisation. The cortical excitability will be measured before and immediately after homeostatic plasticity induction (time point 0-min), and then every 10 minutes for 30 minutes.

Homeostatic plasticity will be induced using tDCS applied to the left primary motor cortex for 7 minutes, followed by a break of 3 minutes and another 5 minutes of tDCS. A constant current of 1mA will be transmitted through the tDCS system (Starstim 32, Neuroelectrics, Barcelona, Spain) using two gelled electrodes placed into holes of a neoprene cap at the position of C3 and Fp2.

The distribution of the data will be tested using a Shapiro-Wilk's test of normality. To investigate the effect of immobilisation and exercise on homeostatic plasticity, a two-way repeated measures analysis of variance (RM-ANOVA) will be conducted with factors Session (Session 1, session 2, and session 3) and Time (baseline, 0 min, 10 min, 20min, and 30 min) and a P value of <0.05 will be considered statistically significant. Adjustments will be made for multiple post-hoc comparisons using appropriate corrections.

ELIGIBILITY:
Inclusion Criteria:

o Healthy, aged between 18-60 years, right-handed, and can speak, read, and understand Danish or English

Exclusion Criteria:

* Pregnant or breastfeeding
* Regular use of cannabis, opioids or other drugs (except contraceptives)
* Current or previous neurologic, musculoskeletal, mental, or other illnesses (e.g. brain or spinal cord injuries, degenerative neurological disorders, epilepsy, major depression, cardiovascular disease, chronic lung disease, etc.)
* Current or previous chronic or recurrent pain condition
* Current regular use of analgesic medication or other medication which may affect the trial (including paracetamol and NSAIDs)
* Lack of ability to cooperate
* Recent history of acute pain particularly in the lower limbs (unless related to low back pain in patients included in sub-project 6)
* Abnormally disrupted sleep in 24 hours preceding experiment
* Any medical or other condition (i.e. musculoskeletal, cardiorespiratory, neurological, etc.)
* Contraindications to TMS application (history of epilepsy, metal implants in head or jaw, etc.)
* Unable to pass the "Transcranial Magnetic Stimulation Adult Safety Screen" or tDCS screening questionnaire

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Corticospinal excitability | Immediately after [0 minutes after homeostatic plasticity induction] and every 10 minutes up until 30 minutes after [10-30 minutes after homeostatic plasticity induction]
  Change in corticospinal excitability (compared to baseline), as reflected by motor-evoked potential amplitudes induced by transcranial magnetic stimulation, after homeostatic plasticity induction

SECONDARY OUTCOMES:
Quantitative Sensory Testing: Cuff detection threshold | Before and 30 minutes post homeostatic plasticity induction
  Cuff detection threshold [kPa]
Quantitative Sensory Testing: Cuff pain tolerance threshold | Before and 30 minutes post homeostatic plasticity induction
  Cuff pain tolerance threshold [kPa]
Quantitative Sensory Testing: Conditioned pain modulation | Before and 30 minutes post homeostatic plasticity induction
  Conditioned pain modulation [kPa change]
Quantitative Sensory Testing: Temporal summation of pain | Before and 30 minutes post homeostatic plasticity induction
  Temporal summation of pain [pain rating; Visual analogue scale; 0-10 cm; higher scores means more pain]
Quantitative Sensory Testing: Mechanical pain threshold | Before and 30 minutes post homeostatic plasticity induction
  Mechanical pain threshold (pin prick) [force required for inducing pricking pain; nM]
Quantitative Sensory Testing: Handheld algometry at right dorsal interosseous muscle | Before and 30 minutes post homeostatic plasticity induction
  Handheld algometry at right dorsal interosseous muscle [kPa]
Quantitative Sensory Testing: Handheld algometry at left dorsal interosseous muscle | Before and 30 minutes post homeostatic plasticity induction
  Handheld algometry at left dorsal interosseous muscle [kPa]
Quantitative Sensory Testing: Handheld algometry at right tibialis anterior muscle | Before and 30 minutes post homeostatic plasticity induction
  Handheld algometry at right tibialis anterior muscle [kPa]
Questionnaires: Pittsburgh Sleep Quality Index | Before baseline corticospinal excitability measurements
  Pittsburgh Sleep Quality Index (PSQI; 0-21; PSQI > 5 means poor sleep quality)
Questionnaires: Pain Catastrophizing Scale | Before baseline corticospinal excitability measurements
  Pain Catastrophizing Scale (PCS; 0-52; higher score means more pain catastrophizing)
Questionnaires: International Physical Activity Questionnaire | Before baseline corticospinal excitability measurements
  International Physical Activity Questionnaire (IPAQ; resting metabolic rate multiplied by activity per minutes performed > higher means better physical activity)
Questionnaires: Positive and Negative Affective Schedule | Before baseline corticospinal excitability measurements
  Positive and Negative Affective Schedule - Short Form (PANAS; 10-50; higher scores = higher levels of negative or positive affect)

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fricke K, Seeber AA, Thirugnanasambandam N, Paulus W, Nitsche MA, Rothwell JC. Time course of the induction of homeostatic plasticity generated by repeated transcranial direct current stimulation of the human motor cortex. J Neurophysiol. 2011 Mar;105(3):1141-9. doi: 10.1152/jn.00608.2009. Epub 2010 Dec 22. PMID 21177994
- [Background] Thapa T, Graven-Nielsen T, Chipchase LS, Schabrun SM. Disruption of cortical synaptic homeostasis in individuals with chronic low back pain. Clin Neurophysiol. 2018 May;129(5):1090-1096. doi: 10.1016/j.clinph.2018.01.060. Epub 2018 Feb 9. PMID 29472134
- [Background] Thapa T, Graven-Nielsen T, Schabrun SM. Aberrant plasticity in musculoskeletal pain: a failure of homeostatic control? Exp Brain Res. 2021 Apr;239(4):1317-1326. doi: 10.1007/s00221-021-06062-3. Epub 2021 Feb 26. PMID 33635391
- [Background] Wittkopf PG, Larsen DB, Gregoret L, Graven-Nielsen T. Prolonged corticomotor homeostatic plasticity - Effects of different protocols and their reliability. Brain Stimul. 2021 Mar-Apr;14(2):327-329. doi: 10.1016/j.brs.2021.01.017. Epub 2021 Jan 24. No abstract available. PMID 33503491